CLINICAL TRIAL: NCT05600231
Title: Twelve Week Clinical Efficacy of Virtually Supervised Mouth Rinse and Flossing: Effect on Plaque, Gingivitis, and Microbiome
Brief Title: A Study of Virtually Supervised Mouth Rinses and Flossing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCSORC004913; CCSORC004913 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Healthy
MeSH Terms: interventions — Ethanol; Mouthwashes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment Group: Brush Only (Experimental): Participants will brush their teeth using a marketed soft bristled toothbrush and Colgate Cavity Protection Toothpaste for 1 timed minute under virtual supervision once daily during the week. At home, participants will brush a second time unsupervised daily in the evening and twice daily over weekends and holidays for 12 weeks. First product use will occur at the site under supervision.
  Interventions: Other: Colgate Cavity Protection Toothpaste
- Treatment Group: Brush / Rinse (LISTERINE COOL MINT Antiseptic Mouthwash) (Experimental): Participants will brush their teeth using a marketed soft bristled toothbrush and Colgate Cavity Protection Toothpaste once daily for 1 timed minute during the week under supervision and rinse with 20 milliliters (mL) of LISTERINE COOL MINT Antiseptic Mouthwash for 30 seconds. At home, participants will brush and rinse a second time unsupervised daily in the evening and twice daily over weekends and holidays for 12 weeks. First product use will occur at the site under supervision.
  Interventions: Other: LISTERINE COOL MINT Antiseptic Mouthwash; Other: Colgate Cavity Protection Toothpaste
- Treatment Group: Brush / Rinse LISTERINE COOL MINT ZERO Alcohol Mouthwash) (Experimental): Participants will brush their teeth using a marketed soft bristled toothbrush and Colgate Cavity Protection Toothpaste once daily for 1 timed minute during the week under supervision and rinse with 20 mL of LISTERINE COOL MINT ZERO Alcohol Mouthwash for 30 seconds. At home, participants will brush and rinse a second time unsupervised daily in the evening and twice daily over weekends and holidays for 12 weeks. First product use will occur at the site under supervision.
  Interventions: Other: LISTERINE COOL MINT ZERO Alcohol Mouthwash; Other: Colgate Cavity Protection Toothpaste
- Treatment Group: Brush / Floss (Experimental): Participants will brush their teeth using marketed soft bristled toothbrush and Colgate Cavity Protection Toothpaste for 1 timed minute and floss with Reach Unflavored Waxed Dental Floss under virtual supervision once daily during the week. At home, participants will brush a second time unsupervised daily in the evening. Over weekends and holidays, participants will brush and floss once daily. Only brushing will be performed a second time in the evening for 12 weeks. First product use will occur at the site under supervision.
  Interventions: Other: Reach Unflavored Waxed Dental Floss; Other: Colgate Cavity Protection Toothpaste
- Treatment Group: Brush / Floss / Rinse (LISTERINE COOL MINT ZERO Alcohol Mouthwash) (Experimental): Participants will brush their teeth using marketed soft bristled toothbrush and Colgate Cavity Protection Toothpaste for 1 timed minute, floss with Reach Unflavored Waxed Dental Floss and rinse with LISTERINE COOL MINT ZERO Alcohol Mouthwash for 30 seconds under virtual supervision once daily during the week. At home, participants will brush and rinse a second time unsupervised daily in the evening. Over weekends and holidays, participants will brush, floss and rinse once daily. Only brushing and rinsing will be performed a second time in the evening for 12 weeks. First product use will occur at the site under supervision.
  Interventions: Other: LISTERINE COOL MINT ZERO Alcohol Mouthwash; Other: Reach Unflavored Waxed Dental Floss; Other: Colgate Cavity Protection Toothpaste
- Healthy Reference Group (No Intervention): Healthy participants will enroll in this reference group and will not receive any study product nor will they receive a prophylaxis as part of their participation in this study. The healthy reference group will be used as a comparator group for microbiome.

INTERVENTIONS:
Other: LISTERINE COOL MINT Antiseptic Mouthwash — Participants will use LISTERINE COOL MINT Antiseptic Mouthwash for 30 second after brushing teeth twice daily.
  Arms: Treatment Group: Brush / Rinse (LISTERINE COOL MINT Antiseptic Mouthwash)
Other: LISTERINE COOL MINT ZERO Alcohol Mouthwash — Participants will use LISTERINE COOL MINT ZERO Alcohol Mouthwash for 30 second after brushing teeth twice daily.
  Arms: Treatment Group: Brush / Floss / Rinse (LISTERINE COOL MINT ZERO Alcohol Mouthwash); Treatment Group: Brush / Rinse LISTERINE COOL MINT ZERO Alcohol Mouthwash)
Other: Reach Unflavored Waxed Dental Floss — Participants after brushing for 1 timed minute, will rinse mouth with water and Floss once a day.
  Arms: Treatment Group: Brush / Floss; Treatment Group: Brush / Floss / Rinse (LISTERINE COOL MINT ZERO Alcohol Mouthwash)
Other: Colgate Cavity Protection Toothpaste — Participants will use Colgate Cavity Protection Toothpaste for brushing teeth twice daily.
  Arms: Treatment Group: Brush / Floss; Treatment Group: Brush / Floss / Rinse (LISTERINE COOL MINT ZERO Alcohol Mouthwash); Treatment Group: Brush / Rinse (LISTERINE COOL MINT Antiseptic Mouthwash); Treatment Group: Brush / Rinse LISTERINE COOL MINT ZERO Alcohol Mouthwash); Treatment Group: Brush Only

SUMMARY:
The purpose of this study is to evaluate the efficacy of brushing, flossing, and rinsing with essential oil mouth rinses; brushing and flossing; versus brushing and rinsing with essential oil mouth rinses; and brushing only for the prevention and reduction of plaque and gingivitis.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and follow the requirements and restrictions of the study (including willingness to use the assigned study products per instructions, availability on scheduled visit dates and likeliness of completing the clinical study) based upon research site personnel's assessment
* Evidence of a personally signed and dated informed consent document indicating the participants has been informed of all pertinent aspects of the trial
* Able to read and understand (participants capable of reading the documents)
* Able to schedule once daily virtual session during weekdays for flossing and rinsing in real time via a platform such as Zoom, Facetime, Google Meet, etc
* Adequate oral hygiene (that is, brush teeth daily and exhibit no signs of oral neglect)
* Adults 18 years of age or older, in good general and oral health without any known allergy to commercial dental products or cosmetics
* Evidence of being fully vaccinated for coronavirus disease-2019 (COVID-19) (adults 60 years and older)
* Negative pregnancy urine tests (females of childbearing potential only)
* Females of childbearing potential must be using a medically-acceptable method of birth control for at least one month prior to visit 1 and agree to continue using this method during their participation in the study
* A minimum of 20 natural teeth with scorable facial and lingual surfaces. Teeth that are grossly carious, extensively restored, orthodontically banded, abutments, exhibiting severe generalized cervical and/or enamel abrasion, or third molars will not be included in the tooth count
* A mean gingival index less than or equal to (<=) 0.75 per the Modified Gingival Index at baseline (healthy reference group)
* A minimum of 10 percent (%) bleeding sites based on the Expanded Bleeding Index (EBI) (randomized treatment groups)
* Participants will have evidence of some gingivitis (mild to severe); there will be no minimum or maximum mean Modified Gingival Index (MGI) score for gingivitis or Turesky Modification of the Quigley Hein Plaque Index (TPI) score for plaque (randomized treatment groups)
* No more than 3 sites having pocket depths of 5 mm and no sites that are greater than 5 millimeters (mm) in depth (randomized treatment groups)
* Absence of significant oral soft tissue pathology, excluding plaque-induced gingivitis, based on a visual examination and at the discretion of the Investigator
* Absence of advanced periodontitis based on a clinical examination and discretion of the dental examiner
* Absence of fixed or removable orthodontic appliance or removable partial dentures or other appliances which may interfere with flossing

Exclusion Criteria:

* History of significant adverse effects, including sensitivities or suspected allergies, following use of oral hygiene products such as toothpastes, mouth rinses and red food dye; Known allergy or sensitivity or history of significant adverse effects to any of the investigational product and/or product ingredients (or other ingredients in the products)
* Dental prophylaxis within four weeks prior to screening/baseline visit
* History of medical conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures
* More than or equal to 3% bleeding sites at baseline (healthy reference group)
* Teeth having periodontal pocket depths measuring more than 3mm in depth (healthy reference group)
* Use of antibiotics, anti-inflammatory or anticoagulant therapy during the study or within the one month prior to the baseline exam. Intermittent use of certain anti-inflammatory medication is acceptable at the discretion of the investigator
* Use of chemotherapeutic anti-plaque/anti-gingivitis products such as triclosan, essential oils, cetylpyridinium chloride, stannous fluoride or chlorhexidine containing mouth rinses and toothpastes within four weeks prior to the baseline
* Regular consumption of probiotic drinks/supplements within one week prior to screening/baseline
* Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results)
* Self-reported smokeless tobacco user including snuff, chewing tobacco, vaping and e-cigarette usage
* Suspected alcohol or substance abuse (example, amphetamines, benzodiazepines, cocaine, marijuana, opiates)
* Significant unstable or uncontrolled medical condition which may interfere with a participant's participation in the study, including cancer, chronic kidney disease, chronic obstructive pulmonary disease (COPD), immunocompromised state (weakened immune system) from solid organ transplant, serious heart conditions, (such as heart failure, coronary artery disease, or cardiomyopathies) sickle cell disease, Type 1 or 2 diabetes mellitus
* Participation in any clinical trial within 30 days of the screening/baseline exam
* Participants who were previously screened and ineligible or were randomized to receive investigational product
* Participants who are related to those persons involved directly or indirectly with the conduct of this study (that is, principal investigator, sub-investigators, study coordinators, other site personnel, employees of Johnson & Johnson subsidiaries, contractors of Johnson & Johnson, and the families of each)
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the participant inappropriate for entry into this study
* COVID-19 restrictions: Participants who fail to meet the criteria of the site's screening consent for preventing Infection in the site's COVID-19 consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Interproximal Mean Turesky Plaque Index (TPI) After 12 Weeks of Product Use | After 12 weeks
  Interproximal Mean TPI after 12 weeks of product use will be reported. Plaque area will be scored by the Turesky Modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (no plaque); 1 (separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (thin, up to 1 millimeter [mm]), continuous band of plaque at the gingival margin); 3 (band of plaque wider than 1mm but less than1/3 of the surface); 4 (plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (plaque covering 2/3 or more of the surface).
Interproximal Mean Modified Gingival Index (MGI) After 12 Weeks of Product Use | After 12 weeks
  Interproximal Mean MGI after 12 weeks of product use will be reported. Gingivitis will be assessed by the Modified Gingival Index on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (normal [absence of inflammation]), 1 (mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (mild inflammation of the entire gingival unit); 3 (moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).

SECONDARY OUTCOMES:
Marginal Mean TPI After 4 and 12 Weeks | After 4 and 12 weeks
  Marginal mean TPI after 4 and 12 weeks will be reported. Plaque area will be scored by the Turesky Modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (no plaque); 1 (separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (thin up to 1 mm), continuous band of plaque at the gingival margin); 3 (band of plaque wider than 1mm but less than1/3 of the surface); 4 (plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (plaque covering 2/3 or more of the surface).
Marginal Mean MGI After 4 and 12 Weeks | After 4 and 12 weeks
  Marginal mean MGI after 4 and 12 weeks will be reported. Gingivitis will be assessed by the Modified Gingival Index on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (normal [absence of inflammation]), 1 (mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (mild inflammation of the entire gingival unit); 3 (moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).
Marginal Mean Expanded Bleeding Index (EBI) After 4 and 12 Weeks | After 4 and 12 weeks
  Marginal mean EBI after 4 and 12 weeks will be reported. Bleeding will be assessed according to the EBI, 168 Sites. A periodontal probe with a 0.5 millimeter (mm) diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degree, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (absence of bleeding after 30 seconds); 1 (bleeding after 30 seconds); 2 (immediate bleeding).
Interproximal Mean TPI After 4 Weeks | After 4 weeks
  Interproximal mean TPI After 4 weeks will be reported. Plaque area will be scored by the Turesky Modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (no plaque); 1 (separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (thin up to 1 mm), continuous band of plaque at the gingival margin); 3 (band of plaque wider than 1mm but less than1/3 of the surface); 4 (plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (plaque covering 2/3 or more of the surface).
Interproximal Mean MGI After 4 Weeks | 4 weeks
  Interproximal mean MGI space after 4 weeks will be reported. Gingivitis will be assessed by the Modified Gingival Index on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (normal [absence of inflammation]), 1 (mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (mild inflammation of the entire gingival unit); 3 (moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).
Whole Mouth Mean TPI After 4 and 12 weeks | After 4 and 12 weeks
  Whole mouth mean TPI after 4 and 12 weeks will be reported. Plaque area will be scored by the Turesky Modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (no plaque); 1 (separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (thin, up to 1 mm), continuous band of plaque at the gingival margin); 3 (band of plaque wider than 1mm but less than1/3 of the surface); 4 (plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (plaque covering 2/3 or more of the surface).
Whole Mouth Mean MGI After 4 and 12 Weeks | After 4 and 12 weeks
  Whole mouth mean MGI after 4 and 12 weeks will be reported. Gingivitis will be assessed by the Modified Gingival Index on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (normal [absence of inflammation]), 1 (mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (mild inflammation of the entire gingival unit); 3 (moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).
Whole Mouth and Interproximal Mean EBI After 4 and 12 Weeks | After 4 and 12 weeks
  Whole mouth and interproximal mean EBI After 4 and 12 Weeks will be reported. Bleeding will be assessed according to the Expanded Gingival Bleeding Index, 168 Sites. A periodontal probe with a 0.5 mm diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degree, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (absence of bleeding after 30 seconds); 1 (bleeding after 30 seconds); 2 (immediate bleeding).
Whole Mouth and Interproximal Percent Bleeding Sites After 4 and 12 Weeks based on EBI | After 4 and 12 weeks
  Whole mouth and interproximal percent bleeding sites after 4 and 12 Weeks based on EBI will be reported. Percent bleeding sites will be calculated by taking the total number of sites with bleeding score greater than 0 divided by the total number of sites assessed for each participant. Bleeding will be assessed according to the Expanded Gingival Bleeding Index, 168 Sites. A periodontal probe with a 0.5 mm diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degree, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (absence of bleeding after 30 seconds); 1 (bleeding after 30 seconds); 2 (immediate bleeding).
Whole Mouth and Interproximal Mean Pocket Depth After 12 Weeks | After 12 weeks
  Whole mouth and interproximal mean pocket depth after 12 weeks will be reported.
Whole Mouth and Interproximal Mean Bleeding Upon Probing Pocket Depths After 12 Weeks | After 12 weeks
  Whole mouth and interproximal mean bleeding upon probing pocket depths after 12 weeks will be reported.
Shannon-Weaver Diversity Index | At baseline and 4 and 12 weeks
  The Shannon-Weaver diversity index will be reported for supragingival plaque assessment.
Total Species Microbial Load | At baseline and 4 and 12 weeks
  The total species microbial load will be reported for supragingival plaque assessment.
Categorical Species Microbial Load | At baseline and 4 and 12 weeks
  The categorical species microbial load will be reported for supragingival plaque assessment.
Bacterial Species Richness | At baseline and 4 and 12 weeks
  The observed bacterial species richness will be reported for supragingival plaque assessment.
Changes in Microbiome Composition by Multidimensional Reduction Analysis | At baseline and 4 and 12 weeks
  Weighted UniFrac principal coordinates analysis (PCoA) analysis for the assessment of microbiome composition shift.
Number of Live Bacterial Counts Expressed in Log10 | Up to 12 weeks
  Quantification of live total bacteria and select species of interest in supragingival plaque using viability quantitative polymerase chain reaction (qPCR) and reported in Log10 bacterial cell number.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Milleman, DDS, Principal Investigator — Salus Research, Inc.
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Bauroth K, Charles CH, Mankodi SM, Simmons K, Zhao Q, Kumar LD. The efficacy of an essential oil antiseptic mouthrinse vs. dental floss in controlling interproximal gingivitis: a comparative study. J Am Dent Assoc. 2003 Mar;134(3):359-65. doi: 10.14219/jada.archive.2003.0167. PMID 12699051
- [Background] Sharma N, Charles CH, Lynch MC, Qaqish J, McGuire JA, Galustians JG, Kumar LD. Adjunctive benefit of an essential oil-containing mouthrinse in reducing plaque and gingivitis in patients who brush and floss regularly: a six-month study. J Am Dent Assoc. 2004 Apr;135(4):496-504. doi: 10.14219/jada.archive.2004.0217. PMID 15127875
- [Background] Sharma NC, Charles CH, Qaqish JG, Galustians HJ, Zhao Q, Kumar LD. Comparative effectiveness of an essential oil mouthrinse and dental floss in controlling interproximal gingivitis and plaque. Am J Dent. 2002 Dec;15(6):351-5. PMID 12691269
- [Background] Newman, MG, Takei, H, Klokkevold, PR, Carranza, FA; 2018; Newman and Carranza's Clinical Periodontology E-Book, 13th Edition; Saunders; p.387.
- [Background] Rich SK, Friedman JA, Schultz LA. Effects of flossing on plaque and gingivitis in third grade schoolchildren. J Public Health Dent. 1989 Spring;49(2):73-7. doi: 10.1111/j.1752-7325.1989.tb02029.x. PMID 2709366
- [Background] Van der Weijden GA, Timmerman MF, Nijboer A, Reijerse E, Van der Velden U. Comparison of different approaches to assess bleeding on probing as indicators of gingivitis. J Clin Periodontol. 1994 Oct;21(9):589-94. doi: 10.1111/j.1600-051x.1994.tb00748.x. PMID 7806674
- [Background] Saxton CA, van der Ouderaa FJ. The effect of a dentifrice containing zinc citrate and Triclosan on developing gingivitis. J Periodontal Res. 1989 Jan;24(1):75-80. doi: 10.1111/j.1600-0765.1989.tb00860.x. PMID 2524573
- [Background] CHILTON NW. Studies in the design and analysis of dental experiments. II. A four-way analysis of variance. J Dent Res. 1960 Mar-Apr;39:344-60. doi: 10.1177/00220345600390021601. No abstract available. PMID 13809868
- [Background] Lobene RR, Weatherford T, Ross NM, Lamm RA, Menaker L. A modified gingival index for use in clinical trials. Clin Prev Dent. 1986 Jan-Feb;8(1):3-6. No abstract available. PMID 3485495
- [Background] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376
- [Derived] Min K, Bosma ML, John G, McGuire JA, DelSasso A, Milleman J, Milleman KR. Quantitative analysis of the effects of brushing, flossing, and mouthrinsing on supragingival and subgingival plaque microbiota: 12-week clinical trial. BMC Oral Health. 2024 May 17;24(1):575. doi: 10.1186/s12903-024-04362-y. PMID 38760758
- [Derived] Bosma ML, McGuire JA, DelSasso A, Milleman J, Milleman K. Efficacy of flossing and mouth rinsing regimens on plaque and gingivitis: a randomized clinical trial. BMC Oral Health. 2024 Feb 3;24(1):178. doi: 10.1186/s12903-024-03924-4. PMID 38310236
- See also: Twelve Week Clinical Efficacy of Virtually Supervised Mouth Rinse and Flossing: Effect on Plaque, Gingivitis, and Microbiome — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSORC004913&attachmentIdentifier=fbbb1940-2e3a-49cb-b218-7fe805c9e7e1&fileName=Floss_Zero_CCSORC004913_Clinical_Study_Report_Redacted_Synopsis_for_ClinTrials.gov_scanned.pdf&versionIdentifier=